CLINICAL TRIAL: NCT06367192
Title: School Readiness Intervention for Preschool Children With Sickle Cell Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SKITS2; K23HL166697 (NIH)
Record Dates: First submitted 2024-04-05; First posted 2024-04-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Readiness Intervention (Experimental): * Attend virtual classroom program sessions- If participants are in the school readiness group, the caregiver, will attend about 8 weeks of sessions virtually with a teacher or social worker and a caregiver of a child with sickle cell, for a total of 8 sessions. The sessions will be during the summer and done in a group. Each session will last about 1 ½ hours and will be video recorded. > •Complete a caregiver interview-If participants are in the school readiness group, a member of the study team will interview you after the virtual classroom sessions are over. The interview will take about 15-20 minutes and will be audio recorded. Participants will be asked for suggestions and how satisfied you were with the program.
  * Complete assessments - Caregiver and participant will complete a set of assessments that evaluate school readiness skills (e.g., early math and reading), child behaviors, and parent-child relationships before and after the intervention.
  Interventions: Behavioral: The adapted Kids in Transition to School Intervention
- Control: Standard school resources (Other): Parents will be provided with information about preschool programs available in the community and age appropriate books for their children
  Interventions: Behavioral: Standard school resources

INTERVENTIONS:
Behavioral: The adapted Kids in Transition to School Intervention — An intensive, school readiness intervention designed to improve preschoolers' social skills, early literacy, numeracy, and self-regulation skills at high risk for academic difficulties. The intervention is delivered virtually over 8 weeks with caregivers and intentionally occurs over the summer when there is a gap in preschool services.
  Other Names: Kids in Transition to School (KITS)
  Arms: Readiness Intervention
Behavioral: Standard school resources — Information about local preschool programs and age appropriate books for children will be provided.
  Arms: Control: Standard school resources

SUMMARY:
The study participant is being asked to take part in this clinical trial, a type of research study, because the participant is a young child with sickle cell disease or the caregiver of a child with sickle cell disease. This study is being done to test a school readiness program for children with sickle cell disease (ages 3.5-6,5 years old).

Primary Objective

Assess feasibility and acceptability of an adapted school readiness intervention among preschool children (ages 3.5-6.5) diagnosed with sickle cell disease.

Secondary Objectives

Objective 1:

Measure preliminary efficacy of the adapted school readiness intervention compared to routine care among preschool children ages (3.5-6.5) diagnosed with sickle cell disease.

Objective 2:

Examine implementation factors (i.e., barriers and facilitators) during post-intervention.

DETAILED DESCRIPTION:
* Group randomization- Parent and child will be randomly selected (like the flip of a coin) to receive either the school readiness intervention or the standard school resources.
* Attend virtual classroom program sessions- If the participant is in the school readiness group, the caregiver, will attend about 8 weeks of sessions virtually with a teacher and a caregiver of a child with sickle cell, for a total of 8 sessions. The sessions will be during the summer and done in a group. Each session will last about 1 ½ hours and will be video recorded. These sessions will be shared with another researcher for feedback and consistency.
* Complete a caregiver interview-If you are in the school readiness group, a member of the study team will interview you after the virtual classroom sessions are over. The interview will take about 15-20 minutes and will be audio recorded. The caregiver will be asked for suggestions and how satisfied with the program.
* Complete assessments - Caregiver and child will complete a set of assessments that evaluate school readiness skills (e.g., early math and reading), child behaviors, and parent-child relationships before and after the intervention.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with sickle cell disease of any genotype.
* Enrolled on the institutional protocol: Sickle Cell Clinical Research Intervention Program (SCCRIP)
* Age 3.5-6.5 years inclusive at the time of enrollment
* English as the primary language
* Research participant and one parent willing to participate and provide consent/assent according to institutional guidelines

Caregiver Participants

* Have a child diagnosed with SCD of any genotype between the ages of 3.5-6.5 years and enrolled in SCCRIP
* English as the primary language

Exclusion Criteria

* Do not have a child diagnosed with SCD of any genotype between the ages of 3.5-6.5 years and enrolled in SCCRIP
* Non-English speakers

Ages: 42 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure | Collected immediately after the intervention
  A brief (4-items) Likert-scale questionnaire assessing feasibility of the intervention. This measure is completed by care givers and intervention providers.
Acceptability of Intervention Measure | Collected immediately after the intervention
  A brief (4-items) Likert-scale questionnaire assessing acceptability of the intervention. This measure is completed by care givers and intervention providers.

SECONDARY OUTCOMES:
Bracken School Readiness Assessment - 3rd Edition | Baseline and Collected immediately after the intervention
  A Standardized assessment of school readiness skills for preschool children.
Woodcock Johnson Tests of Achievement - Fourth Edition | Baseline and Collected immediately after the intervention
  A standardized measure of reading, mathematics, and spelling.
NIH Toolbox Flanker Test | Baseline and Collected immediately after the intervention
  A computerized test of inhibitory control.
Head-Toes-Knees-Shoulders Revised | Baseline and Collected immediately after the intervention
  A behavioral measure that examines self-regulation in preschool children.
Behavior Rating Inventory of Executive Functioning Preschool or Child | Baseline and Collected immediately after the intervention
  A parent rating form that assesses executive functioning using a set of standardized questions.
The Parenting Scale | Baseline and Collected immediately after the intervention
  A self-report measure completed by caregivers assessing their parenting skills.

CONTACTS AND LOCATIONS:
Overall Officials: ANDREW Heitzer, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols